CLINICAL TRIAL: NCT06913179
Title: CAR-T Cell Therapy Combined With Allogeneic Hematopoietic Stem Cell Transplantation for Relapsed/Refractory Multiple Myeloma
Brief Title: CAR-T Cell Therapy Combined With Allogeneic Hematopoietic Stem Cell Transplantation for Relapsed or Refractory Multiple Myeloma
Acronym: CAR-T-allo
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Kai Lin Xu，MD, Pro., Xuzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2025-KL061-01; XYFY2025-KL061-01 (Other: The Affiliated Hospital oh Xuzhou Medical University)
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- allo-HSCT following CAR-T (Experimental): All enrolled patients will first receive CAR-T cell therapy. Patients who achieve complete remission (CR) following CAR-T infusion will subsequently undergo allogeneic hematopoietic stem cell transplantation (allo-HSCT) based on clinical assessment. The entire treatment process will be standardized and closely monitored, with follow-up evaluations focusing on adverse events, engraftment success, relapse risk, and overall survival.
  Interventions: Biological: All enrolled patients will first receive CAR-T cell therapy. Patients who achieve complete remission following CAR-T infusion will subsequently undergo allo-HSCT

INTERVENTIONS:
Biological: All enrolled patients will first receive CAR-T cell therapy. Patients who achieve complete remission following CAR-T infusion will subsequently undergo allo-HSCT — All enrolled patients will first receive CAR-T cell therapy. Patients who achieve complete remission (CR) following CAR-T infusion will subsequently undergo allogeneic hematopoietic stem cell transplantation (allo-HSCT) based on clinical assessment. The entire treatment process will be standardized and closely monitored, with follow-up evaluations focusing on adverse events, engraftment success, relapse risk, and overall survival.

SUMMARY:
1. Study Title CAR-T Cell Therapy Combined with Allogeneic Hematopoietic Stem Cell Transplantation for Relapsed or Refractory Multiple Myeloma
2. Study Objective This study aims to evaluate the safety and efficacy of CAR-T cell therapy followed by allogeneic hematopoietic stem cell transplantation (allo-HSCT) in patients with relapsed or refractory multiple myeloma. The goal is to explore a novel treatment strategy for this high-risk patient population.
3. Study Design This is a single-center, open-label, single-arm clinical study. A total of 30 patients with relapsed or refractory multiple myeloma will be enrolled. All participants will receive standardized CAR-T cell therapy followed by allo-HSCT and will undergo systematic observation and follow-up to assess therapeutic efficacy and safety.
4. Sample Size A total of 30 patients will be enrolled in this study.
5. Eligibility Criteria (1) Inclusion Criteria Age between 18 and 70 years; Estimated life expectancy of more than 12 weeks; Diagnosis of multiple myeloma confirmed by physical examination, pathology, laboratory tests, and imaging studies; Patients with refractory multiple myeloma; Patients with relapsed multiple myeloma; ALT and AST < 3 times the upper limit of normal; Total bilirubin < 2.0 mg/dL; Karnofsky Performance Status (KPS) > 50%; No severe dysfunction of major organs such as liver, kidney, or heart; Prior failure of autologous or allogeneic hematopoietic stem cell transplantation; Ineligible for stem cell transplantation or patients who declined transplantation due to other constraints; Voluntarily willing to receive CAR-T cell therapy for B cell-derived hematologic malignancies; Suitable for peripheral venous blood collection with no contraindications to leukapheresis; Able to understand and sign a written informed consent form.

(2) Exclusion Criteria Pregnant or lactating women, or women planning pregnancy within 6 months; Presence of infectious diseases (e.g., HIV infection, active tuberculosis); Active hepatitis B or C virus infection; Pre-screening indicates peripheral blood T-cell transduction efficiency < 10% or expansion fold < 5× under CD3/CD28 co-stimulation; Abnormal vital signs or inability to cooperate with treatment procedures; Presence of psychiatric or psychological disorders that affect treatment compliance or outcome assessment; History of severe allergy or hypersensitivity, particularly to interleukin-2 (IL-2); Systemic or localized severe infections requiring anti-infective therapy; Significant dysfunction of critical organs such as heart, lung, brain, or kidney; Patients with severe autoimmune diseases; Any other conditions deemed unsuitable for enrollment by the investigator.

6. Treatment Protocol All enrolled patients will first receive CAR-T cell therapy. Patients who achieve complete remission (CR) following CAR-T infusion will subsequently undergo allogeneic hematopoietic stem cell transplantation (allo-HSCT) based on clinical assessment. The entire treatment process will be standardized and closely monitored, with follow-up evaluations focusing on adverse events, engraftment success, relapse risk, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 70 years; Estimated life expectancy of more than 12 weeks; Diagnosis of multiple myeloma confirmed by physical examination, pathology, laboratory tests, and imaging studies; Patients with refractory multiple myeloma; Patients with relapsed multiple myeloma; ALT and AST < 3 times the upper limit of normal; Total bilirubin < 2.0 mg/dL; Karnofsky Performance Status (KPS) > 50%; No severe dysfunction of major organs such as liver, kidney, or heart; Prior failure of autologous or allogeneic hematopoietic stem cell transplantation; Ineligible for stem cell transplantation or patients who declined transplantation due to other constraints; Voluntarily willing to receive CAR-T cell therapy for B cell-derived hematologic malignancies; Suitable for peripheral venous blood collection with no contraindications to leukapheresis; Able to understand and sign a written informed consent form.

Exclusion Criteria:

Pregnant or lactating women, or women planning pregnancy within 6 months; Presence of infectious diseases (e.g., HIV infection, active tuberculosis); Active hepatitis B or C virus infection; Pre-screening indicates peripheral blood T-cell transduction efficiency < 10% or expansion fold < 5× under CD3/CD28 co-stimulation; Abnormal vital signs or inability to cooperate with treatment procedures; Presence of psychiatric or psychological disorders that affect treatment compliance or outcome assessment; History of severe allergy or hypersensitivity, particularly to interleukin-2 (IL-2); Systemic or localized severe infections requiring anti-infective therapy; Significant dysfunction of critical organs such as heart, lung, brain, or kidney; Patients with severe autoimmune diseases; Any other conditions deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Month 6, 12, 18 and 24
  The proportion of patients achieving partial response (PR) or better according to the IMWG criteria.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Month 6, 12, 18 and 24
  Time from CAR-T infusion to disease progression or death from any cause.
Overall Survival (OS) | Month 6, 12, 18 and 24
  Time from CAR-T infusion to death from any cause.

IPD SHARING:
Plan to Share IPD: No